CLINICAL TRIAL: NCT06202066
Title: A Phase II Study of Temozolomide and Survivin Long Peptide Vaccine (SurVaxM) in Patients With Progressing Metastatic Neuroendocrine Carcinomas (NECs)
Brief Title: Temozolomide and Survivin Long Peptide Vaccine (SurVaxM) for the Treatment of Patients With Progressing Metastatic Neuroendocrine Carcinomas
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: pending protocol changes
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 3622923; NCI-2023-09345 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 3622923 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Digestive System Neuroendocrine Neoplasm; Lung Neuroendocrine Neoplasm; Malignant Solid Neoplasm; Pancreatic Neuroendocrine Neoplasm
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Specimen Handling; montanide ISA 51; incomplete Freund's adjuvant; Magnetic Resonance Spectroscopy; sargramostim; Colony-Stimulating Factors; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- (temozolomide, SurVaxM) (Experimental): Patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity and can be continued at investigators discretion at end of treatment. Patients also receive SurVaxM with montanide ISA-51 SC and sargramostim SC once every 2 weeks for 4 doses. Patients with clinical benefit after 4 doses of SurVaxM and remain free of tumor progression and unacceptable toxicity may receive 3 additional doses on weeks 24, 36, and 48. Additionally, patients undergo blood sample collection, CT scans or MRI scans throughout study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Incomplete Freund''s Adjuvant; Procedure: Magnetic Resonance Imaging; Biological: Sargramostim; Biological: SVN53-67/M57-KLH Peptide Vaccine; Drug: Temozolomide

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Incomplete Freund''s Adjuvant — Given SC
  Other Names: Freund's Incomplete Adjuvant; IFA; incomplete Freund's adjuvant; ISA-51; Montanide ISA 51; Montanide ISA-51
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: SVN53-67/M57-KLH Peptide Vaccine — Given SC
  Other Names: SurVaxM
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase IIa trial compares the safety and effect of temozolomide combined with survivin long peptide vaccine (SurVaxM) to temozolomide alone in patients with neuroendocrine tumors (NET) that has spread from where it first started (primary site) to other places in the body (metastatic) and is growing, spreading or getting worse (progressing). Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid and may kill tumor cells and slow down or stop tumor growth. Survivin, a protein, is expressed in 50% of patients that have neuroendocrine tumors and, is associated with poor outcomes. SVN53-67/M57-KLH peptide vaccine (SurVaxM) is a vaccine that has been shown to produce an immune system response against cancer cells that express a survivin and may block the growth of new tumor cells. Giving temozolomide with SurVaxM may kill more tumor cells in patients with progressing metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To determine the clinical efficacy (progression free survival [PFS]) of combining temozolomide and SVN53-67/M57-KLH peptide vaccine (SurVaxM) in patients with progressing NECs.
* To evaluate the safety and toxicity of the study drug combination (temozolomide + SurVaxM) in patients with progressing NECs.

SECONDARY OBJECTIVES:

I. To assess clinical benefit (including complete response, partial response and stable disease as defined by Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1) at 3 months, 6 months, 9 months, and 12 months from study entry.

II. To assess anti-survivin IgG titer response.

EXPLORATORY OBJECTIVES:

I. To explore immune markers associated with clinical responses to SurVaxM in peripheral blood of NETs patients.

II. To assess the methylguanine methyltransferase (MGMT) status of all patients and correlate with response.

III. To assess the tumor growth rate (TGR) on radiographic imaging prior to study enrollment and while on study.

OUTLINE:

Patients receive temozolomide orally (PO) once daily (QD) on days 1-5. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity and can be continued at investigators discretion at end of treatment. Patients also receive SurVaxM with incomplete Freund's adjuvant (montanide ISA-51) subcutaneously (SC) and sargramostim SC once every 2 weeks for 4 doses. Patients with clinical benefit after 4 doses of SurVaxM and remain free of tumor progression and unacceptable toxicity may receive 3 additional doses on weeks 24, 36, and 48. Additionally, patients undergo blood sample collection, computed tomography (CT) scans or magnetic resonance imaging (MRI) scans throughout study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Have a Karnofsky performance status ≥ 80 or Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (i.e. the patient must be able to care for himself/ herself with occasional help from others)
* Measurable, pathologically confirmed diagnosis of neuroendocrine tumor of gastrointestinal, pancreatic, or lung origin with ki67>20% or neuroendocrine carcinoma of any origin excluding small cell lung carcinoma (well-differentiated G3 NETs and extrapulmonary NECs).
* Patients must have documented radiographic progression, determined as clinically significant by the treating provider, within the last twelve months on two CT or MRI scans performed at least four weeks apart per RECIST v1.1 criteria. In the case of retreatment, progression may be defined by the treating provider (e.g., clinical, radiographic, biochemical)
* Patients must have failed at least one prior systemic therapy
* Patients who have been on somatostatin analogues (SSA) may continue to take SSA while on study treatment
* Archival neuroendocrine tumor tissue must test positive for survivin presence by clinical immunohistochemistry prior to study enrollment
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (obtained within 14 days prior to enrollment)
* Platelets ≥ 100 x 10^9/L (obtained within 14 days prior to enrollment)
* Hemoglobin (Hgb) > 9g/dL (obtained within 14 days prior to enrollment)
* Plasma total bilirubin: ≤ 1.5 x upper limit of normal (ULN) (obtained within 14 days prior to enrollment)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 4 x ULN (obtained within 14 days prior to enrollment)
* Creatinine clearance ≥ 60 mL/min (per Cockroft-Gault equation) (obtained within 14 days prior to enrollment)
* Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight [LMW] heparin) must meet the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices, which carries a significant risk of bleeding in investigator's opinion)
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have received temozolomide in the advanced disease setting either alone or as part of a combination therapy will be excluded if they progressed while on it
* Has received prior treatment with SurVaxM
* Received an investigational agent within 30 days prior to enrollment
* Participants who have received checkpoint inhibitors within 3 months prior to study enrollment or, those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, bradycardia, tachycardia or psychiatric illness/social situations that would limit compliance with study requirements and, which in the treating physicians' opinion would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for at least 3 years are eligible for this study
* Known history of an autoimmune disorder
* Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness
* Systemic corticosteroid therapy > 2mg of dexamethasone or equivalent per day at study entry
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Patients with Hepatitis B or Hepatitis C may be included if there are adequately controlled viral titers and no drug-drug interactions, testing not required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | At 6 months
  Summarized using frequencies and relative frequencies.
Incidence of adverse events | Up to 1 year
  Defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse events (CTCAE) version (v) 5.0. Adverse events will be summarized by attribution and grade using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Response | At 3, 6, 9 and 12 months from study entry
  Assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Response will be summarized by time-point using frequencies and relative frequencies. Clinical benefit (best response of complete response [CR], partial response [PR] or stable disease [SD]) will be estimated and summarized using frequencies and relative frequencies, with a 95% confidence interval obtained for the clinical benefit rate.
Overall survival (OS) | At the time from treatment initiation until death due to any cause up to 1 year
  OS will be summarized using standard Kaplan-Meier methods, where the median will be estimated with a 95% confidence interval.
Time to progression (TTP) | At the time from treatment initiation until disease progression, death or last follow up up to 1 year
  Defined using RECIST v1.1. TTP will be summarized using standard Kaplan-Meier methods, where the median will be estimated with a 95% confidence interval.
Titer response | Up to 1 year
  Defined as anti-survivin IgG titers > 30,000 and will be summarized using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Renuka V Iyer, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States